CLINICAL TRIAL: NCT00524342
Title: Phase II Clinical Efficacy Trial of Recombinant Interleukin-11 (rhIL-11, Neumega) in Women With Type 1 Von Willebrand Disease and Refractory Menorrhagia
Brief Title: IL-11 in Women With Von Willebrand Disease and Refractory Menorrhagia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Margaret Ragni (Other)
Collaborators: University of North Carolina (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Margaret Ragni, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO07040157; Wyeth 102344 (Other: Wyeth)
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Von Willebrand Disease
Keywords: IL-11; von Willebrand disease; von Willebrand factor; VWFmRNA; menorrhagia
MeSH Terms: conditions — von Willebrand Diseases; Menorrhagia | interventions — oprelvekin; Interleukin-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oprelvekin, Interleukin 11, IL-11 (Experimental): 25 micrograms/kg by subcutaneous injection once daily for four days, then once daily on day 1-7 during each of six consecutive menstrual cycles
  Interventions: Drug: Oprelvekin, Interleukin 11, IL-11

INTERVENTIONS:
Drug: Oprelvekin, Interleukin 11, IL-11 — 25 micrograms/kg by subcutaneous injection once daily for four days, then once daily on day 1-7 during each of six consecutive menstrual cycles
  Other Names: Neumega (Oprelvekin, Interleukin 11, IL-11)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of rhIL-11, when given subcutaneously for six consecutive months, in reducing menstrual blood loss in women with type 1 von Willebrand disease and refractory menorrhagia. Efficacy will be measured by subjective bleeding severity scale and pictorial bleeding chart. Safety will be measured by the frequency of adverse events, including fever, headache, fatigue, myalgias, arthralgias, fluid retention, or edema.

DETAILED DESCRIPTION:
This study is a prospective, single-center Phase II trial of Neumega (rhIL-11) in women with type 1 VWD and menorrhagia refractory to estrogen, hormones, or hemostatic agents. It is anticipated that 10 subjects who meet eligibility criteria will enroll and complete this study. All aspects of this study, including the rhIL-11 injections and the screening, hemostatic and safety monitoring, and coagulation testing, are considered experimental. The specific objectives are to determine the efficacy and safety of rhIL-11 in reducing menstrual blood loss in adult women with type 1 VWD during six consecutive menstrual cycles, and to determine the mechanism of the hemostatic response of rhIL-11.

ELIGIBILITY:
Inclusion Criteria:

* Females 18-45 years of age
* Confirmed type 1 VWD, as defined by low VWF:RCoF or low VWF:Ag and qualitatively normal VWF multimers
* Menorrhagia refractory to estrogens, hormones, hemostatic agents
* Willingness to have blood drawn

Exclusion Criteria:

* Use of immunomodulatory or experimental drugs, or diuretics
* Pregnant or lactating women or those unwilling to use contraception during study
* Previous cardiac disease, congestive failure, arrhythmia (e.g., atrial fibrillation, atrial flutter), hypertension, MI, stroke, or thrombosis
* Past allergic reaction to Neumega or DDAVP
* Surgery within the past 8 weeks
* Inability to comply with study protocol requirements
* Concomitant use of antiplatelet drugs, anticoagulants, dextran, aspirin or NSAIDs
* Treatment with DDAVP, cryoprecipitate, whole blood, plasma and plasma derivatives containing substantial quantities of FVIII and/or VWF within five days of study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret V. Ragni, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hemophilia Center of Western PA, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Jankowitz RC, Nichols TC, Ragni MV. Recombinant IL-11 (Neumega, rhIL-11) increases plasma Von Willebrand Factor in Type 1 Von Willebrand Disease. Blood 108: 1003, 2006 (abstract).
- [Background] Ragni MV, Jankowitz RC, Chapman HL, Merricks EP, Kloos MT, Dillow AM, Nichols TC. A phase II prospective open-label escalating dose trial of recombinant interleukin-11 in mild von Willebrand disease. Haemophilia. 2008 Sep;14(5):968-77. doi: 10.1111/j.1365-2516.2008.01827.x. Epub 2008 Aug 1. PMID 18680527
- [Result] Ragni MV, Jankowitz RC, Jaworski K, Merricks EP, Kloos MT, Nichols TC. Phase II prospective open-label trial of recombinant interleukin-11 in women with mild von Willebrand disease and refractory menorrhagia. Thromb Haemost. 2011 Oct;106(4):641-5. doi: 10.1160/TH11-04-0274. Epub 2011 Aug 11. PMID 21833452

RESULTS

PARTICIPANT FLOW:
Groups:
- IL-11: Neumega (Oprelvekin, Interleukin 11, IL-11): 25 micrograms/kg by subcutaneous injection once daily for four days, then once daily on day 1-7 during each of six consecutive menstrual cycles
Period: Overall Study
Arm/Group | IL-11
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IL-11
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: >50% Reduction in PBAC (Pictorial Blood Assessment Chart) at 6 Months
Description: Subjective estimate of blood loss was measured by using a Pictorial blood assessment chart (PBAC) . The PBAC measures scores on a scale where 0 to 100 is normal and greater than 100-200 are abnormal.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | IL-11
Number analyzed (Participants) | 7
percentage of participants | 71

2. Secondary Outcome: No. of Subjects With Detectable VWF mRNA (Von Willebrand Factor Messenger RNA).
Description: No. of subjects with detectable VWFmRNA, a measure of IL-11 (interleukin-11) function, specifically increasing VWF synthesis.
Time Frame: The time frame is up to 7 months per subject.
Measure: Number; unit: participants
Arm/Group | IL-11
Number analyzed (Participants) | 7
participants | 7

3. Secondary Outcome: No. of Subjects With IL-11 Associated Adverse Events.
Description: The number of subjects with IL-11 associated adverse events.
Time Frame: The time frame is up to 7 months per subject.
Measure: Number; unit: participants
Arm/Group | IL-11
Number analyzed (Participants) | 7
participants
  fluid retention | 6
  injection site bruising | 6
  flushing | 3

ADVERSE EVENTS:
Time Frame: up to 7 months
Arm/Group | IL-11
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IL-11 (N=7)
conjunctival erythema (Skin and subcutaneous tissue disorders) | 7
fluid retention (General disorders) | 6
injection site bruising (General disorders) | 6
flushing (General disorders) | 3
thrombocytosis (Blood and lymphatic system disorders) | 1
hypokalemia (Renal and urinary disorders) | 1
diastolic hypertension (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes